CLINICAL TRIAL: NCT01339845
Title: Introduction of Cholera Vaccine in Bangladesh: " Impact Evaluation of Cholera Vaccine and Behaviour Change Interventions in Urban Dhaka"
Brief Title: Introduction of Cholera Vaccine in Bangladesh
Acronym: ICVB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Directorate General of Health Services, Ministry of Health and Family Welfare, Bangladesh (Unknown); International Vaccine Institute (Other); Dhaka City Corporation, Ministry of Local Government and Rural Development, Bangladesh (Unknown); School of Public Health and Health Professions, University at Buffalo, USA (Unknown); Johns Hopkins Bloomberg School of Public Health (Other); University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PR-10061
Record Dates: First submitted 2011-04-01; First posted 2011-04-21 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-02

CONDITIONS: Cholera
Keywords: Cholera vaccine; Behaviour change intervention; Cost effectiveness and cost-benefit; Prevention of cholera; Control of Cholera; Vaccination
MeSH Terms: conditions — Cholera | interventions — shanchol; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vaccine arm (Active Comparator): Thirty clusters (approximately 80,000 people) will receive cholera vaccine alone
  Interventions: Biological: ShanChol
- Vaccine plus hygiene and safe water arm (Active Comparator): Thirty clusters (approximately 80,000 people)will receive both cholera vaccine and behaviour change
  Interventions: Behavioral: Vaccine and behaviour
- Non-intervention arm (No Intervention): 30 neighbourhoods(approximately 80,000 people) will continue their standard habits and practices

INTERVENTIONS:
Biological: ShanChol — Each dose of the vaccine contains whole cell Killed inactivated V.cholerae O1 and O139 strains.Vaccine is packaged as liquid formulations in 1.5-ml doses. The vaccine is given two doses separated by a two week interval and administered orally.
  Arms: Vaccine arm
Behavioral: Vaccine and behaviour — Together with vaccination the community health worker will offer a hand washing station and water treatment facilities that include both hardware and a software component. The idea of the handwashing station is to bring together with soap and water that people need for handwashing, especially for handwashing after defecation. The hardware for water treatment is a chlorine dispenser that is a reservoir which holds sodium hypochlorite and dispenses a measured dose of the dilute sodium hypochlorite into a 15 liter water tank. Community residents can collect water directly from the 15 L water tanks into their own personal water storage vessels. The community health worker will negotiate with compound residents for the development of a water treatment system.
  Arms: Vaccine plus hygiene and safe water arm

SUMMARY:
The purpose of this study is to conduct and evaluate the feasibility and effectiveness of a mass cholera vaccination program to reduce diarrhea due to Vibrio cholerae in a high incidence urban area. This study will also evaluate the feasibility of adding a household hand washing and safe drinking water promotion intervention to a cholera vaccine program and the overall impact of this combination on decreasing the incidence of diarrhea due to Vibrio cholerae.

DETAILED DESCRIPTION:
Cholera continues to be a major cause of morbidity and mortality in low income countries including Bangladesh. It is estimated that there are at least 300,000 severe cases and 1.2 million infections in people in Bangladesh each year. Deaths annually from cholera may have decreased but overall morbidity remains high.

The project for "Introduction of Cholera Vaccine in Bangladesh" (ICVB) will examine the effectiveness of intervention with an oral cholera vaccine in reducing incidence of cholera in urban Dhaka, and the effectiveness of a handwashing and home water treatment behaviour change intervention in reducing diarrhea due to cholera. The proposal involves evaluation of a 2-dose regimen of an oral killed whole cell (WC) vaccine and a handwashing and home water treatment behavior change program promoting improved hygiene and home drinking water treatment in reducing dehydrating diarrhea in a low income area of Dhaka, Bangladesh. The study population will include 90 clusters (neighborhoods) in an area of high cholera incidence in Mirpur with a total study population of 240,000. Thirty clusters (approximately 80,000 people) will receive cholera vaccine alone, 30 clusters will receive both cholera vaccine and behavior change and 30 neighborhoods will continue their standard habits and practices. Surveillance for cholera and diarrhea will be carried out in all the three areas during the whole project period. Following the GIS mapping and census of the target populations, the cholera vaccine will be offered to all males and non-pregnant females aged one year and above in the vaccination areas, and an aggressive hygiene and safe water promotion program will be implemented in the 30 behavior change communication clusters. Passive surveillance for cholera will be undertaken using the two ICDDR,B diarrhea treatment facilities as well as 10 other health facilities that serve the study areas. Vaccine and other public health coverage and costs effectiveness as well cost-benefit will be measured, followed by surveillance and identical follow-up studies. The hygiene and safe water behavior change program will also be continued for 4 years. The impact of interventions will be assessed by following vaccination by directly comparing the incidence of cholera and diarrhea in the intervention communities to the incidence in the standard habits and practices communities.

ELIGIBILITY:
Inclusion Criteria:

1. Apparently healthy residents of selected vaccination sites
2. Aged 1 year and above
3. Non-pregnant women
4. Written informed consent

Exclusion Criteria:

1. Age less than 1 year
2. Pregnant women

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240000 (Actual)
Dates: Start 2009-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of individuals vaccinated with two dose of oral cholera vaccine. | Six months from initiation of vaccination
  Tergated individuals will be vaccinated and vaccination records will give the coverage.
Decrease number of cholera cases in intervention arm compared to non-intervention arm. | Two years after completion of vaccination
  The primary analyses will be comparison of the incidence of primary outcome in the intervention clusters compared to the non-intervention cluster

SECONDARY OUTCOMES:
Incidence of cholera among vaccinated individuals in vaccination area. | Two years after completion of vaccination.
  Vaccine-induced protective immunity will be estimated from comparing the incidence of cholera among vaccine recipients in the vaccination area and the incidence of cholera among vaccine non-recipients in the same area.
Incidence of cholera among non-vaccinated individuals in vaccination area. | Two years after completion of vaccination
  Indirect protection (herd protection), the protection of non-vaccinated persons due to reduced transmission of an infection, will be estimated from comparing the incidence of cholera among non-vaccinees in the vaccination area and the incidence of cholera in the control area.
Incidence of cholera in the combined cholera vaccine and behavior change intervention area | Two years after completion of vaccination
  Assessment of the impact of the combined cholera vaccine and behavior change intervention on the incidence of all diarrheas treated at the ICDDRB and other health facilities.

CONTACTS AND LOCATIONS:
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Dhaka Division, Bangladesh

REFERENCES:
- [Background] Sur D, Lopez AL, Kanungo S, Paisley A, Manna B, Ali M, Niyogi SK, Park JK, Sarkar B, Puri MK, Kim DR, Deen JL, Holmgren J, Carbis R, Rao R, Nguyen TV, Donner A, Ganguly NK, Nair GB, Bhattacharya SK, Clemens JD. Efficacy and safety of a modified killed-whole-cell oral cholera vaccine in India: an interim analysis of a cluster-randomised, double-blind, placebo-controlled trial. Lancet. 2009 Nov 14;374(9702):1694-702. doi: 10.1016/S0140-6736(09)61297-6. Epub 2009 Oct 8. PMID 19819004
- [Background] Mahalanabis D, Lopez AL, Sur D, Deen J, Manna B, Kanungo S, von Seidlein L, Carbis R, Han SH, Shin SH, Attridge S, Rao R, Holmgren J, Clemens J, Bhattacharya SK. A randomized, placebo-controlled trial of the bivalent killed, whole-cell, oral cholera vaccine in adults and children in a cholera endemic area in Kolkata, India. PLoS One. 2008 Jun 4;3(6):e2323. doi: 10.1371/journal.pone.0002323. PMID 18523643
- [Derived] Jefferson T, Dooley L, Ferroni E, Al-Ansary LA, van Driel ML, Bawazeer GA, Jones MA, Hoffmann TC, Clark J, Beller EM, Glasziou PP, Conly JM. Physical interventions to interrupt or reduce the spread of respiratory viruses. Cochrane Database Syst Rev. 2023 Jan 30;1(1):CD006207. doi: 10.1002/14651858.CD006207.pub6. PMID 36715243
- [Derived] Kang S, Chowdhury F, Park J, Ahmed T, Tadesse BT, Islam MT, Kim DR, Im J, Aziz AB, Hoque M, Pak G, Khanam F, Ahmmed F, Liu X, Zaman K, Khan AI, Kim JH, Marks F, Qadri F, Clemens JD. Are better existing WASH practices in urban slums associated with a lower long-term risk of severe cholera? A prospective cohort study with 4 years of follow-up in Mirpur, Bangladesh. BMJ Open. 2022 Sep 21;12(9):e060858. doi: 10.1136/bmjopen-2022-060858. PMID 36130764
- [Derived] Ali M, Qadri F, Kim DR, Islam MT, Im J, Ahmmed F, Khan AI, Zaman K, Marks F, Kim JH, Clemens JD. Effectiveness of a killed whole-cell oral cholera vaccine in Bangladesh: further follow-up of a cluster-randomised trial. Lancet Infect Dis. 2021 Oct;21(10):1407-1414. doi: 10.1016/S1473-3099(20)30781-7. Epub 2021 Jun 16. PMID 34146473
- [Derived] Jefferson T, Del Mar CB, Dooley L, Ferroni E, Al-Ansary LA, Bawazeer GA, van Driel ML, Jones MA, Thorning S, Beller EM, Clark J, Hoffmann TC, Glasziou PP, Conly JM. Physical interventions to interrupt or reduce the spread of respiratory viruses. Cochrane Database Syst Rev. 2020 Nov 20;11(11):CD006207. doi: 10.1002/14651858.CD006207.pub5. PMID 33215698
- [Derived] Saha A, Hayen A, Ali M, Rosewell A, MacIntyre CR, Clemens JD, Qadri F. Socioeconomic drivers of vaccine uptake: An analysis of the data of a geographically defined cluster randomized cholera vaccine trial in Bangladesh. Vaccine. 2018 Jul 25;36(31):4742-4749. doi: 10.1016/j.vaccine.2018.04.084. Epub 2018 May 8. PMID 29752024
- [Derived] Khan AI, Ali M, Chowdhury F, Saha A, Khan IA, Khan A, Akter A, Asaduzzaman M, Islam MT, Kabir A, You YA, Saha NC, Cravioto A, Clemens JD, Qadri F. Safety of the oral cholera vaccine in pregnancy: Retrospective findings from a subgroup following mass vaccination campaign in Dhaka, Bangladesh. Vaccine. 2017 Mar 13;35(11):1538-1543. doi: 10.1016/j.vaccine.2017.01.080. Epub 2017 Feb 11. PMID 28196715
- [Derived] Qadri F, Ali M, Chowdhury F, Khan AI, Saha A, Khan IA, Begum YA, Bhuiyan TR, Chowdhury MI, Uddin MJ, Khan JAM, Chowdhury AI, Rahman A, Siddique SA, Asaduzzaman M, Akter A, Khan A, Ae You Y, Siddik AU, Saha NC, Kabir A, Riaz BK, Biswas SK, Begum F, Unicomb L, Luby SP, Cravioto A, Clemens JD. Feasibility and effectiveness of oral cholera vaccine in an urban endemic setting in Bangladesh: a cluster randomised open-label trial. Lancet. 2015 Oct 3;386(10001):1362-1371. doi: 10.1016/S0140-6736(15)61140-0. Epub 2015 Jul 9. PMID 26164097
- [Derived] Khan IA, Saha A, Chowdhury F, Khan AI, Uddin MJ, Begum YA, Riaz BK, Islam S, Ali M, Luby SP, Clemens JD, Cravioto A, Qadri F. Coverage and cost of a large oral cholera vaccination program in a high-risk cholera endemic urban population in Dhaka, Bangladesh. Vaccine. 2013 Dec 9;31(51):6058-64. doi: 10.1016/j.vaccine.2013.10.021. Epub 2013 Oct 22. PMID 24161413